CLINICAL TRIAL: NCT02539940
Title: A Prospective Observational Study Using Elutax-SV Drug-eluting Balloons for Below-the-knee Treatment
Brief Title: Elutax-SV Drug-eluting Balloons for Below-the-knee Treatment
Acronym: Apollo
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: Zentrum für Klinische Studien Jena (Other); Aachen Resonance GmbH (Industry)
Responsible Party: Principal Investigator, Ulf Teichgräber, Prof. Dr. med., Jena University Hospital
Other Study IDs: 4448-06/15
Record Dates: First submitted 2015-08-17; First posted 2015-09-03 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Critical Limb Ischemia; Peripheral Artery Disease
Keywords: Below-the-knee
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with critical limb ischemia: Patients undergoing endovascular intervention of below-the-knee arteries with ELUTAX SV DEB (drug-eluting balloon).
  Interventions: Device: Angioplasty Paclitaxel-eluted balloon catheter ELUTAX SV

INTERVENTIONS:
Device: Angioplasty Paclitaxel-eluted balloon catheter ELUTAX SV — Angioplasty for revascularization in below-the-knee arteries

SUMMARY:
The aim of this observational study is to evaluate the outcomes and safety of the Paclitaxel-eluted balloon catheter ELUTAX SV for treatment of peripheral arterial disease (PAD) in below-the-knee vessels

DETAILED DESCRIPTION:
The management of critical limb ischemia due to below-the-knee disease remains challenging due to the frequent patient comorbidities, diffuse vascular involvement, limb preservation, and high rates of restenosis and disease progression. This study will record the use of ELUTAX SV-DEB under real life conditions in a representative sample.The investigators will generate new data in observing the outcome and the safety of the Elutax SV drug-eluting balloons for change in Rutherford clinical category from baseline to 6 and 12 month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Paclitaxel-eluting balloon angioplasty in below-the-knee lesions with ELUTAX SV-DEB
* Age ≥ 18 years
* Signed informed consent
* documented Critical Limb Ischemia (CLI) in the target limb prior to the study
* Rutherford Category 4, 5 or 6
* ≥70% diameter stenosis or occlusion in the target lesion, including de-novo / in-stent restenosis/occlusion of target lesion
* Patent inflow artery
* Target vessel(s) diameter between 2 and 4 mm
* Target vessel(s) reconstitute(s) at or above the ankle

Exclusion Criteria:

* Life expectancy below 50% within the next 12 months (as judged by the investigator)
* Planned major index limb amputation
* Acute limb ischemia (within last 14 days thrombectomy, atherectomy, or lysis)
* Application of DEB-eluting balloons except from ELUTAX SV in the same target limb (POBA is allowed)
* Patient unwilling or unlikely to comply with follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients in Germany who undergo treatment with the ELUTAX SV-DEB that is applied for treatment of peripheral arterial disease (PAD) in below-the-knee vessels.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2015-09; Primary Completion 2018-04 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change of Rutherford Classification | after 6 and 12 month
  Change of Rutherford stage to baseline at Follow-up visits

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (10):
  - DRK Kliniken Berlin Köpenick, Berlin, Brandenburg
  - Oberlausitz-Kliniken Bautzen, Bautzen, Saxony
  - Städtisches Krankenhaus Dresden-Friedrichstadt, Dresden, Saxony
  - Heinrich-Braun-Krankenhaus, Zwickau, Saxony
  - Klinikum Altenburger Land GmbH, Altenburg, Thuringia
  - SRH-Waldklinikum, Gera, Thuringia
  - University Hospital Jena, Radiology, Jena, Thuringia
  - Saale-Unstrut Klinikum Naumburg, Naumburg, Thuringia
  - MEDINOS Kliniken Sonneberg, Sonneberg, Thuringia
  - Kreiskrankenhaus Torgau "J. Kentmann" gGmbH, Torgau

REFERENCES:
- [Derived] Teichgraber U, Lehmann T, Thieme M, Wahl KU, Stelzner C, Bormann A, Gotz L, Kroessner T, Boden H, Maiwald L, Aschenbach R. Drug-Coated Balloon Angioplasty of Infrapopliteal Lesions in Patients with Critical Limb Ischaemia: 1-Year Results of the APOLLO Trial. Cardiovasc Intervent Radiol. 2019 Oct;42(10):1380-1390. doi: 10.1007/s00270-019-02279-6. Epub 2019 Jul 8. PMID 31286197